CLINICAL TRIAL: NCT03487055
Title: Safety Assessment of Repeated Administration of a Fully Human Monoclonal Antibody of RNAKL (TK006) in Patients With Breast Cancer-related Bone Metastases
Brief Title: Safety Assessment of Repeated Administration of TK006 in Patients With Breast Cancer-related Bone Metastases
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tmab-TK006-102b
Record Dates: First submitted 2018-03-13; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): The subjects would receive 120 mg TK006 every 4-week over a period of 84 days.
  Interventions: Biological: TK006

INTERVENTIONS:
Biological: TK006 — Subcutaneous injection in the upper arm
  Other Names: fully human monoclonal anti-RANKL antibody

SUMMARY:
This is an open labelled study. It was designed to evaluate the safety of multiple-dosing of TK006 in patients with breast cancer-related bone metastases. This trial is the extension of a core study: Phase 1 Trial of a Fully Human Monoclonal Antibody of Receptor Activator for Nuclear Factor-κ B Ligand (RNAKL, TK006) Safety, Pharmacokinetics, and Pharmacodynamics in Patients With Breast Cancer-related Bone Metastases (NCT 03239756).

DETAILED DESCRIPTION:
This trial is the extension of a core study: Phase 1 Trial of a Fully Human Monoclonal Antibody of Receptor Activator for Nuclear Factor-κ B Ligand (RNAKL, TK006) Safety, Pharmacokinetics, and Pharmacodynamics in Patients With Breast Cancer-related Bone Metastases (NCT 03239756). It's an open labelled study, aimed at evaluating the safety of repeated administration of TK006 in patients with breast cancer-related bone metastases. The qualified subjects would be those completed the entire observation in either 60 mg, 120 mg or 180 mg single dose arm at the core study. Also, these patients should be well-tolerated with TK006 at the core study and are deemed to further benefit from this extension phase estimated by the researcher and sponsor. The subjects would receive 120 mg TK006 every 4-week over a period of 84 days.

Only safety profile and immunogenicity assessment would be assessed in this extension stage, and no further study on pharmacokinetics and pharmacodynamics would be done.

ELIGIBILITY:
Inclusion Criteria:

1. Patients provide written informed consent voluntarily.
2. 18~65 years old, male or female.
3. Patients who completed the entire observation in either 60 mg, 120 mg or 180 mg single dose arm at the core phase (NCT 03239756). Also, these patients should be well-tolerated with TK006 and would further benefit from continued treatment estimated by the researcher and sponsor.
4. ECOG≤2.
5. Albumin-adjusted calcium≥2.0mmol/L, ≤2.9mmol/ L.

Exclusion Criteria:

1. Women in pregnancy or nursing.
2. Central nervous system metastasis that is symptomatic or require treatment.
3. Patients with grade III or IV adverse events considered related to TK006 at the core phase (NCT 03239756).
4. Patients with important organs dysfunction and not suitable for further treatment with TK006 judged by the researcher.
5. Imaging confirmed progression in bone metastasis compared with core phase (NCT 03239756).
6. Previous or existing osteomyelitis or osteonecrosis of jaw, toothache or jaw diseases which are in active or require invasive operations, unhealed wound of oral surgery, or planned invasive dental operations during this trial.
7. Patients who have been selected for the study of other test devices or test medicine.
8. Other situations which are not suitable for participation judged by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events（AEs）which are related to TK006 treatment throughout the study | 85 days
  Adverse events refer to any treatment related abnormality with clinical significance identified by means of vital signs examination, physical check-up, twelve leads electrocardiogram inspection and laboratory tests throughout the study. Adverse events reported by subjects would also be recorded in the entire trial. All these abnormal cases described above would be reported as incidence of adverse events.

SECONDARY OUTCOMES:
immunogenicity | 85 days
  Neutralization antibody of TK006 would be detected on the day 0 (before dosing), day 28 (before dosing) and day 84.

CONTACTS AND LOCATIONS:
Overall Officials: jiang H Y, Study Director — Jiangsu T-Mab Biopharma Co.,Ltd